CLINICAL TRIAL: NCT02699541
Title: The Effectiveness of Information-Motivation-Behavioural Skills Model-based Diabetes Self-Management Education Among Patients With Type 2 Diabetes in Jordan
Brief Title: The Effectiveness of Diabetes Self-Management Education Program Based on Behavioural Change Theory
Acronym: IMB-DSME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14946
Record Dates: First submitted 2016-02-17; First posted 2016-03-04 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Health Behavior; Diabetes Mellitus, Type 2
Keywords: Diabetes Self-Management Education; Behavioural change theory; IMB model; Diabetes Type 2
MeSH Terms: conditions — Health Behavior; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intervention group participants will receive the educational intervention based on the Information, Motivational, Behavioral change model.
  Interventions: Behavioral: Diabetes Self-Management Education
- Control group (No Intervention): Control group participants will receive usual care treatment and referral to diabetes educational consultation if required.

INTERVENTIONS:
Behavioral: Diabetes Self-Management Education — This study will implement an individualized DSME program based on Information-Motivation-Behavioral (IMB) skills theory. IMB behavioral change theory assumption proposes that health-related behavior information, motivation and behavioural skills are primary determinants of promoting health behavior.
  Researcher will use a previously validated educational toolkit (PRIDE) and will be delivered using motivational interviewing techniques through several sessions for each participant. Two face-to-face sessions (one at the beginning and one at the end of the 3 month period) and one phone call per week or per fortnight.
  Arms: Intervention group

SUMMARY:
In this study, researchers will test the effectiveness of a self-management education programme, on self-management behaviours of patients with type two diabetes. Up to 230 consenting participants will be recruited from outpatient diabetes clinics in Jordan, 230 participants will be randomised to one of two groups. Group 1 ( 115 patients) have received the intervention, which consisted of an introductory session of tailored, face-to-face education and advice, followed by educational materials to take away, and regular telephone support at a regularity specified by the patient, over a three-month period. This intervention is based on behavioural change theory called the Information-Motivational-Behavioural skills model. Group 2 (115 patients) have received usual clinical care with no additional intervention. Researchers have assessed the effectiveness of the intervention by measuring self-care strategies (dietary habits, physical activity and managing diabetes medications), diabetes control (HbA1c), quality of life and Diabetes Self-Management Knowledge, Motivation and Self-Efficacy at 3 time points: before the intervention, at 3 months and at 6 months.

DETAILED DESCRIPTION:
Background: Type 2 Diabetes (T2DM) is prevalent, costly to healthcare services and associated with significant mortality; over 1.5 million deaths occur directly by diabetes in low and middle-income countries (WHO,2014) and diabetes is predicted to be the seventh leading cause of death by 2030. Ajlouni et al (2008) estimated that approximately one million people in Jordan have been diagnosed with type 2 diabetes; a figure that is increasing. More than half a million Jordanians have an uncontrolled level of Glycosylated Hemoglobin (HbA1c >7.5%) due to factors such as sedentary lifestyle and poor medication management. To prevent diabetes microvascular and macro vascular complications, increased efforts and attention need to be directed towards improving glycaemic levels and improving metabolic outcomes through appropriate glycaemic management. Intensive diabetes management by anti-hyperglycaemic medications alone may improve metabolic outcomes, but may also lead to side effects for patients such as hypoglycaemia and weight gain. Patients with diabetes are strongly recommended to engage in self-management over their glucose levels and this may be best achieved through educating patients in self-management of diabetes.

Didactic interventions have shown to improve metabolic outcomes, although benefits last less than six months and are not sustained in the long term. Educational programs need to target psychological factors such as patient's confidence, to ensure self-management strategies are sustained in the long term. Barriers in diabetes self-management behaviours map on to the Information-Motivation-Behavioural skills (IMB) Model of behavioural change. The model was critically constructed based on analysing previous interventions and addressing limitations of the theories that have been used among clients with HIV risk. Chang et al (2014) systematically reviewed the IMB model-based behavioural interventions and found that effects of IMB model persisted up to 12 months in studies followed up patients for 12 months.

Aim: To examine the effects of IMB Model-based Diabetes Self-Management Educational (DSME) intervention on three self-management activities: patients' eating habits, physical activity and medications management, in patients who attend an outpatients diabetes clinics at Jordan University Hospital and Prince Hamzeh Hospital in Jordan. The hypothesis to be tested is that the IMB educational program will improve participants' behavioural outcomes in self-care at 6 months compared with control participants.

Research protocol and methods: A two group trial with randomised allocation of 230 participants on 1:1 average for both groups. Intervention group will receive the educational intervention. Control group will receive usual clinical care and referral to diabetes educational consultation if required. This intervention is an individualised DSME program based on Information-Motivation-Behavioural (IMB) skills theory. IMB behavioural change theory assumption proposes that health-related behaviour information, motivation and behavioural skills are primary determinants of promoting health behaviour. The intervention will be based on a validated DSME toolkit and will be delivered using motivational interviewing techniques through a two face-to-face session and follow-up phone calls at patients preferred frequency for a period of 3 months.

Data collection will occur at 3 time points; baseline, 3 months and 6 months. Measures will include self-management knowledge, motivation, behavioural skills, diabetes outcomes (HbA1c), blood pressure and weight. At 3 months, some participants in the intervention group will be selected using purposive sampling, to participate in a process evaluation interview.

Measurable end point/statistical power of the study: Primary outcome is diabetes self-care activities measured at 6 months using the Summary of Diabetes Self-Care Activities Scale (SDSCA) questionnaire. Statistical power of 0.8 has been used to calculate study sample.

ELIGIBILITY:
Eligibility criteria:

Patients will be eligible if:

1. They are diagnosed with type 2 DM for more than 6 months to ensure that hyperglycaemia they had experienced was the primary cause of type 2 DM.
2. Attending the clinic regularly once each 3 months for the last two appointments.
3. Taking any form of hypoglycaemic agents (pills or injections such as insulin).

Inclusion criteria:

1. Any age from 18 to 65 years.
2. Access to a telephone whether mobile phone or land line phone (cable).
3. Capable to give informed consent for themselves as well as being able to communicate, read, write and understand Arabic language in order to complete self-report outcomes questionnaires and interpret the study booklet.
4. Experiencing uncontrolled glycaemic level (HbA1c >8%) at the day of visiting the clinic.

Exclusion criteria:

1. Patients who suffer from any cognitive impairment or any disease condition or taking medication that affects their memory (self-reported by patient and/or companion).
2. Pregnant women because they require a specific treatment intervention due to the differences in metabolic outcomes cut off points.
3. Patients who anticipate they will be admitted to the hospital during study period.
4. Currently attending or have attended any diabetes education program in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Participants' diabetes self-Management activities: diet habits, physical activity and medications Management | 6 months
  The primary outcome will be diabetes self-management activities and will be measured by two scales; Summary of Diabetes self-care activities scale (SDSCA) and Medications Adherence Rating Scale (MARS) for each participant.
  Both of them will assess participants' response each by units on a scale, and each participant will have a total score calculated by summing SDSCA score and MARS score.

SECONDARY OUTCOMES:
Participants' glycaemic level. | 6 months
  Glycaemic level will be measured by the (HbA1c) lab test using the percentage unit. A blood test done for each participant each visit during the usual treatment care.
Participants' weight. | 6 months
  Weight will be measured by Kilogram unit using an electric digital scale. Weight is included in the usual physical examination for each participant each visit.
Participants' blood pressure | 6 months
  Blood pressure will be measured by electric device using mm/hg unit. Blood pressure is included in the usual physical examination for each participant each visit.
Participants' quality of life. | 6 months
  Diabetes patients' quality of life will be measured by using Audit of Diabetes Dependent Quality of Life (ADDQoL) by units on a scale score.
Diabetes Self-Management Knowledge | 6 months
  Diabetes Self-Management Knowledge will be measured by using Spoken Knowledge in Low Literacy in Diabetes Scale (SKILLD) by units on a scale score.
Diabetes Self-Management Motivation. | 6 months
  Diabetes Self-Management Motivation will be measured by using both Diabetes Empowerment Scale (DES) + Medical Outcomes Study Social Support Survey (MOS-SSS).
  Both of them will assess participants' response each by units on a scale, and each participant will have a total score calculated by summing DES score and MOS-SSS score.
Diabetes Self-Management Self-Efficacy. | 6 months
  Diabetes Self-Management Self-Efficacy will be measured by using Perceived Diabetes Self-Management Scale (PDSMS).

CONTACTS AND LOCATIONS:
Overall Officials: Holly Blake, PhD, Study Chair — University of Nottingham
Locations (2):
- Jordan (2):
  - Jordan University Hospital, Amman
  - Prince Hamzeh Hospital, Amman

IPD SHARING:
Plan to Share IPD: Undecided